CLINICAL TRIAL: NCT04725149
Title: Investigating the Efficacy of Low or High Dose Tart Cherry on Recovery From Exercise Induced Muscle Damage and Establishing Its Molecular Mechanisms of Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PEP-1905
Record Dates: First submitted 2021-01-20; First posted 2021-01-26 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Muscle Recovery
Keywords: cherry; tart cherry; Montmorency cherry; beverage; exercise; muscle recovery; muscle soreness; muscle damage; muscle function; muscle strength; muscle biopsy; mechanism; oxidative stress; inflammation; anthocyanin; polyphenol; antioxidant; cyclo-oxygenase; myotube; mygenic culture
MeSH Terms: conditions — Motor Activity; Myalgia; Inflammation | interventions — Water

STUDY DESIGN:
Intervention Model Description: Repeated measures, double-blind, counter-balanced
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Taste-matched placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0 ml tart cherry concentrate (Placebo Comparator): Still cherry-flavored beverage, similar in appearance, taste, aroma and calories to the 30 ml and 60 ml tart cherry concentrate beverages
  Interventions: Other: 500 ml base solution
- 30 ml tart cherry concentrate (Experimental): "Low dose" tart cherry concentrate beverage
  Interventions: Other: 500 ml containing 30 ml tart cherry concentrate diluted with water and base solution
- 60 ml tart cherry concentrate (Experimental): "High dose" tart cherry concentrate beverage
  Interventions: Other: 500 ml containing 60 ml tart cherry concentrate diluted with water only

INTERVENTIONS:
Other: 500 ml base solution — Color, taste, aroma, and calorie matched water base
  Arms: 0 ml tart cherry concentrate
Other: 500 ml containing 30 ml tart cherry concentrate diluted with water and base solution — Montmorency cherry concentrate
  Arms: 30 ml tart cherry concentrate
Other: 500 ml containing 60 ml tart cherry concentrate diluted with water only — Montmorency cherry concentrate
  Arms: 60 ml tart cherry concentrate

SUMMARY:
To determine the dose-response effects of 10-day tart cherry product consumption (0, 30 ml, and 60 ml) on knee extensor isometric strength 24-h and 48-h after muscle damaging exercise and to elucidate the mechanisms of action for TC supplementation.

DETAILED DESCRIPTION:
Montmorency cherry supplementation has been shown to exert antioxidant and anti-inflammatory effects that can be beneficial for improving recovery from exercise. However, the investigator is currently not aware of how tart cherry polyphenol supplementation produces these effects. This study aims to determine the dose-response effects of 10-day tart cherry product consumption (placebo, 30 ml, and 60 ml Montmorency tart cherry concentrate in a 500 ml beverage) on knee extensor isometric strength 24-h and 48-h after muscle damaging exercise on supplementation Day 8; on enhancing recovery of other measures of muscle function (single leg eccentric and concentric force development and single leg jump height) and muscle soreness; on reducing markers of oxidative stress and inflammation in plasma, muscle and urine; on inducing signaling in muscle via the nuclear factor erythroid 2-related factor 2 (Nrf2) pathway to upregulate endogenous antioxidant enzymes in muscle; on inhibiting muscle cyclo-oxygenase (COX-1 and COX-2).

This study also aims to identify and establish the molecular mechanisms of action through which tart cherry polyphenols exert antioxidant and anti-inflammatory effects. Oxidative stress and inflammatory signaling in primary human myogenic cells will be assessed by incubating primary human myogenic cells (commercial cell line) in sera derived from 6 participants consuming 8-day placebo vs. 60 ml/day Montmorency tart cherry concentrate supplement. Subjects are permitted to participate in both the molecular mechanism of action part of the study (Part A, no exercise component) and the damaging exercise muscle recovery part of the study (Part B).

For 60 ml doses in Parts A and B, global proteomics analysis of the muscle tissue will be conducted generate more insight into the mechanisms of action. This would identify the specific pathways that are influenced by cherry supplementation and allow identification of the full range of mechanisms involved, rather than assume antioxidant/anti-inflammatory effects alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male in good health
2. 18-40y
3. BMI ≤ 29.9
4. Recreationally active but not highly trained (Participating in sport or physical activity at least once per week for the last 6 months and lower limb resistance training ≤ 1/week) (Part B only)
5. No lower limb musculoskeletal injury that prevented exercise in the last 3 months (Part B only)
6. Understanding of the procedures to be undertaken as part of the study
7. Willing to participate in the exercise protocols (Part B only) and follow supplementation guidelines and other instructions provided by the experimenter
8. Willing to abstain from caffeine, alcohol and strenuous exercise for two 5 day periods (from 48h prior to muscle damaging exercise and throughout the follow up period; days 6-10 of the trial) for Part B, and abstain from caffeine and alcohol for two 3-day periods for Part A
9. Willing to keep food diaries for the duration of each arm of the trial and avoid multiple servings per day of foods that have a high polyphenol content from a list provided.
10. Willing to construct their diet for the first arm of the trial from a list of recipes provided, and to then replicate this diet during the second arm of the trial.
11. Willing to wear a triaxial accelerometer throughout each arm of the trial, and during the second arm of the trial to replicate their physical activity pattern completed in the first arm of the trial.
12. Willing to abstain from consumption of anti-inflammatory, analgesic medications or those with anti-coagulant effects especially NSAIDs and aspirin for 48h prior to and throughout each arm of the trial. (Part B only)
13. Willing to abstain from icing or applying compression bandages to the exercised/biopsied leg (Part B only)
14. Ability to provide voluntary written informed consent to participate in the study.

Exclusion Criteria:

1. Female
2. <18y or >40y
3. BMI ≥ 30
4. Inactive or well-trained (see inclusion criteria) (Part B only)
5. Lower limb musculoskeletal injury in the last 3 months (Part B only)
6. Under the care of a physician
7. Known health condition that could interfere with any element of the data collection protocol. Any known pulmonary, gastrointestinal (e.g., irritable bowel syndrome, Crohn's disease), kidney, cardiovascular, or metabolic diseases, blood-borne infections, or coagulopathies including deep vein thrombosis (DVT)
8. Current regular consumption of nutritional/dietary supplements or previous use of any dietary supplements in the past 6 months known to have a lasting effect.
9. Current use of prescription medication; including the use of an inhaler
10. Non-steroidal anti-inflammatory drugs, aspirin or other analgesic medication or any anti-coagulants are prohibited during the study and for 48h prior to commencing supplementation
11. Allergy/sensitivity/intolerance to cherries, any cherry derived product, or any of the additional ingredients found within the TC test products, including sensitivity to sorbitol.
12. Allergy to lidocaine or other local anaesthetics. (Part B only)
13. Active drug or alcohol dependency
14. Current or active usage of nicotine or tobacco related products
15. Participation in a clinical trial within the past 30 days or concurrently during this trial
16. Participation in any PepsiCo trial within past 6 months, except that Part A participants may take part in Part B after a >=14 day washout from Part A
17. Inability to provide written informed consent

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Isometric knee extensor strength | Changes from immediately before and immediately after muscle damaging exercise on day 8 of tart cherry supplementation to 24 hours and 48 hours after muscle damaging exercise (days 9 and 10 of supplementation).
  Maximum voluntary contraction (MVC) as a measure of functional recovery from muscle damage. Unit of measurement is Newtons. Stronger is better.

SECONDARY OUTCOMES:
Single leg eccentric and concentric isokinetic force production | Changes from immediately before and immediately after muscle damaging exercise on day 8 of tart cherry supplementation to 24 hours and 48 hours after muscle damaging exercise (days 9 and 10 of supplementation).
  Dynamic muscle strength measured by isokinetic contraction (IKC, 60 deg.s-1). More forceful is better.
Single leg vertical jump height (SLVJ) | Changes from immediately before and immediately after muscle damaging exercise on day 8 of tart cherry supplementation to 24 hours and 48 hours after muscle damaging exercise (days 9 and 10 of supplementation).
  Dynamic muscle strength measured by jump height (cm). Higher is better.
Leg muscle soreness by Pressure Pain tolerance (PPT) | Changes from immediately before and immediately after muscle damaging exercise on day 8 of tart cherry supplementation to 24 hours and 48 hours after muscle damaging exercise (days 9 and 10 of supplementation).
  Pressure pain tolerance (PPT) measured by algometer. Higher tolerance is better.
Leg muscle soreness by Visual Analogue Scale (VAS) | Changes from immediately before and immediately after muscle damaging exercise on day 8 of tart cherry supplementation to 24 hours and 48 hours after muscle damaging exercise (days 9 and 10 of supplementation).
  Measured using a visual analogue pain scale from 0 mm (no pain) to 100 mm (extremely painful). Lower score is better.
Leg muscle biopsy for nuclear factor k-B (NFκB) | Changes from pre and post exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Biopsies are done after blood samples and before muscle soreness measures.
  Inflammation marker expression activity of the NFκB pathway will be measured by immunoblotting. Lower is better.
Leg muscle biopsy for cyclo-oxygenase COX1 protein | Changes from pre and post exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Biopsies are done after blood samples and before muscle soreness measures.
  Inflammation marker of cyclo-oxygenase measured by total protein carbonylation (immunoblotting). A reduction (inhibiting) is better.
Leg muscle biopsy for cyclo-oxygenase COX1 activity | Changes from pre and post exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Biopsies are done after blood samples and before muscle soreness measures.
  Inflammation marker of cyclo-oxygenase activity measured by commercially available colorimetric assay. A reduction (inhibiting) is better.
Leg muscle biopsy for nuclear factor erythroid 2-related factor 2 (Nrf2), absolute expression, nuclear translocation | Changes from pre and post muscle damaging exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Biopsies are done after blood samples and before muscle soreness measures.
  Oxidative damage marker Nrf2 pathway intended to upregulate endogenous antioxidant enzymes in muscle. Induction of signaling is better.
Leg muscle biopsy for global proteomics analysis of muscle tissue samples for the 60 ml dose only | Changes from pre and post muscle damaging exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Biopsies are done after blood samples and before muscle soreness measures.
  Tissue analysis to identify pathways influenced by cherry supplementation and identify mechanisms of action.
Leg muscle biopsy for endogenous antioxidant enzyme expression | Changes from pre and post muscle damaging exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Biopsies are done after blood samples and before muscle soreness measures.
  Enzymes (superoxide dismutase 1, superoxide dismutase 2, glutathione peroxidase 1 and catalase) protein expression quantified by immunoblotting. Higher values (upregulation by Nrf2) is better.
Leg muscle biopsy for immune cell infiltration | Changes from pre and post muscle damaging exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Biopsies are done after blood samples and before muscle soreness measures.
  Inflammation marker response measured by immunohistochemistry. Less infiltration is better.
Plasma interleukin-6 (IL-6) | Changes from pre and post muscle damaging exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Pre exercise blood sampling is done after urine collection. Post exercise blood sampling done before biopsy.
  Plasma inflammatory stress response measured by ELISA. A reduction is better.
Plasma protein carbonyls | Changes from pre and post muscle damaging exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Pre exercise blood sampling is done after urine collection. Post exercise blood sampling done before biopsy.
  Oxidative stress response and antioxidant status measured by ELISA. A reduction is better.
Plasma phenolic concentration | Changes from pre and post muscle damaging exercise on day 8 of tart cherry supplementation to pre-exercise on days 9 and 10 of supplementation. Pre exercise blood sampling is done after urine collection. Post exercise blood sampling done before biopsy.
  LC-MS-MS metabolite analysis to evaluate plasma levels associated with tart cherry supplementation at 0, 30 and 60 ml/day.
Urine oxidation-reduction potential (ORP) | Change from pre-exercise value day 8 to days 9 and 10 of tart cherry supplementation. Collected upon arrival to the study site.
  Urinary oxidation-reduction potential to measure oxidative damage and antioxidant status measured by probe. Less oxidative stress/free radical production is better.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Bowtell, PhD, Principal Investigator — University of Exeter, Sport and Health Sciences Department
Locations (1):
- University of Exeter Sport and Health Sciences Department, Exeter, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No